CLINICAL TRIAL: NCT00355238
Title: A Phase II Open Label Study of Brivanib (BMS582664), Administered Orally At A Dose of 800 mg Daily In Subjects With Unresectable, Locally Advanced or Metastatic Hepatocellular Carcinoma Who Have Received Either No Prior Systemic Therapy or One Prior Regimen of Angiogenesis Inhibitor Therapy
Brief Title: A Phase II Open Label Study of BMS-582664 in Locally Advanced or Metastatic Hepatocellular Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA182-006
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — brivanib; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): no comparator to brivanib
  Interventions: Drug: brivanib (active)

INTERVENTIONS:
Drug: brivanib (active) — Tablet, Oral, Brivanib 800 mg, once daily, until progression
  Other Names: BMS-582664

SUMMARY:
The purpose of this clinical research study is to learn if BMS-582664 can shrink or slow the growth of advanced liver cancer. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma (HCC) ≥ 2cm based on:
* Biopsy OR
* Radiological evidence of HCC by contrast-enhanced CT scan or contrast-enhanced AND
* Blood test positive for Hepatitis B or C AND
* Alpha fetoprotein above > 400 mg/L
* Not appropriate for curative surgery
* Screening Blood Pressure <150/100 mmHg, Left Ventricular Ejection Fraction (LVEF) >50%

Exclusion Criteria:

* Heart Attack within 12 months, uncontrolled chest pain within 6 months
* Ascites resistant to diuretic medication therapy
* Portal-systemic encephalopathy
* Portal hypertension with bleeding esophageal or gastric varices within the past 2 months
* Deficiency of sodium in the blood with sodium < 125 mEq/L
* Subjects with serious non-healing wounds, ulcers or bone fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2006-12-31 (Actual); Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (18):
  - City Of Hope National Medical Center, Duarte, California
  - Harbor UCLA Medical Center, Los Angeles, California
  - Harbor-Ucla Medical Center, Los Angeles, California
  - Christiana Care Health Services, Newark, Delaware
  - University Of Miami Miller School Of Medicine, Miami, Florida
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - University Of Chicago, Chicago, Illinois
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - The Cancer Center At Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Univ Of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- France (4):
  - Local Institution, Marseille
  - Local Institution, Reims
  - Local Institution, Rennes
  - Local Institution, Villejuif
- Local Institution, Shatin, Nt.,, Hong Kong
- Malaysia (2):
  - Local Institution, Kampung Baharu Nilai, Negeri Sembilan
  - Local Institution, Kuala Lumpur
- Philippines (3):
  - Local Institution, Cebu City
  - Local Institution, Davao City
  - Local Institution, Quezon
- Local Institution, Singapore, Singapore
- South Korea (2):
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
- Taiwan (2):
  - Local Institution, Tainan
  - Local Institution, Taipei

REFERENCES:
- [Derived] Park JW, Finn RS, Kim JS, Karwal M, Li RK, Ismail F, Thomas M, Harris R, Baudelet C, Walters I, Raoul JL. Phase II, open-label study of brivanib as first-line therapy in patients with advanced hepatocellular carcinoma. Clin Cancer Res. 2011 Apr 1;17(7):1973-83. doi: 10.1158/1078-0432.CCR-10-2011. Epub 2011 Feb 24. PMID 21349999
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort D data collection is not in scope of the planned primary and secondary endpoints per protocol amendment 07.
  Participants who are randomized into the doxorubicin arm and cross-over to brivanib prior to or after this amendment will not be included as treated participants in Arm A, B, or C.
Groups:
- Group A (Brivanib 800 mg QD): Participants with no prior systemic therapy receive brivanib (800 mg) daily (QD).
- Group B (Brivanib 800 mg QD): Participants with one prior regimen of angiogenesis inhibitor therapy treated with brivanib (800 mg) daily (QD).
- Group C (400 mg BID): Participants with one prior regimen of angiogenesis inhibitor therapy treated with brivanib (400 mg) twice daily (BID).
- Cohort D: Doxorubicin: All participants who received at least 1 dose of doxorubicin prior to Protocol Amendment 7. Participants treated with doxorubicin from the original protocol were allowed to cross-over to recieve brivanib alaninate after unequivocal disease progression (no cross-over was allowed for toxicity alone) providing they still met the eligibility criteria and had recovered from doxorubicin toxicities.
Period: Overall Study
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID) | Cohort D: Doxorubicin
Started | 55 | 46 | 22 | 14
Crossed Over From Doxorubicin to Recieve Brivanib Alaninate | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 55 | 46 | 22 | 14
Not completed — Adverse event unrelated to study drug | 2 | 2 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Disease progression | 37 | 36 | 16 | 11
Not completed — Study drug toxicity | 11 | 7 | 5 | 2
Not completed — Participant withdrew consent | 3 | 1 | 0 | 0
Not completed — Participant request to discontinue study treatment | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID) | Cohort D: Doxorubicin | Total
Number analyzed (Participants) | 55 | 46 | 22 | 14 | 137
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 41 | 34 | 13 | 9 | 97
  >= 65 | 14 | 12 | 9 | 5 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 3 | 1 | 23
  Male | 49 | 33 | 19 | 13 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Other | 5 | 3 | 2 | 1 | 11
  Black/ African American | 2 | 3 | 0 | 0 | 5
  Chinese | 11 | 5 | 0 | 1 | 17
  Korean | 18 | 23 | 15 | 7 | 63
  Malaysian | 1 | 0 | 0 | 0 | 1
  White | 18 | 12 | 4 | 5 | 39
  Native Hawaiian/ Other Pacific Islander | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate at 6 Months Per Independent Response Review Committee (IRRC) in Cohort A
Description: The percent of participants who have not progressed or died prior to 6 months from the date of their first dose. Participants who have neither progressed nor died but had their last tumor assessment prior to 6 months will not be categorized as progression free and will not be included. Tumor response was measured by the IRRC using mWHO criteria.
  Progression is defined as a 25% or more increase in the sum of all index lesion areas taking as reference the smallest sum recorded at or following baseline.
Time Frame: From first dose up to approximately 6 months after first dose
Population: All treated participants with no prior systemic therapy (Pre-specified in Group A participants only).
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Group A (Brivanib 800 mg QD)
Number analyzed (Participants) | 55
Percent of participants | 22.4 [10.9 to 33.9]

2. Primary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have to have a causal relationship with this treatment.
Time Frame: From first dose up to 30 days post last dose (up to approximately 34 months)
Population: Pre-specified for all treated participants in group A, B, and C only
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID)
Number analyzed (Participants) | 55 | 46 | 22
Participants | 54 | 46 | 22

3. Secondary Outcome: Tumor Response Rate Per Independent Response Review Committee (IRRC)
Description: The percent of participants whose best overall response is a partial response (PR) or complete response (CR). Tumor measurements by CT/ MRI of the chest, abdomen and pelvis will be obtained at pre-treatment (within 28 days prior to the start of treatment) and every 6 weeks.
  Complete Response (CR): Disappearance of all known disease. Must be confirmed 4 or more weeks later.
  Partial Response (PR): A 50% or more decrease in the sum of all index lesion areas compared to the baseline sum and no unequivocal progression of existing non-index lesions. In addition, there can be no appearance of new lesions. Must be confirmed 4 or more weeks later.
Time Frame: From first dose to the date of the first documented response (up to approximately 34 months)
Population: Pre-specified for all treated participants in group A, B, and C only
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID)
Number analyzed (Participants) | 55 | 46 | 22
Percent of participants | 7.3 [2.0 to 17.6] | 4.3 [0.5 to 14.8] | 0.0 [NA to NA] — Insufficient number of participants with events

4. Secondary Outcome: Disease Control Rate Per Independent Response Review Committee (IRRC)
Description: The percent of participants whose best response is a partial response (PR), complete response (CR) or stable disease (SD).
  Complete Response (CR): Disappearance of all known disease. Must be confirmed 4 or more weeks later.
  Partial Response (PR): A 50% or more decrease in the sum of all index lesion areas compared to the baseline sum and no unequivocal progression of existing non-index lesions. In addition, there can be no appearance of new lesions. Must be confirmed 4 or more weeks later.
  Stable Disease (SD): A decrease of 50% or more or an increase of 25% or more in the sum of all index lesion areas compared to baseline cannot be established. There can be no appearance of new lesions. Documentation must occur 6 weeks (42 days) or more from the baseline determination.
Time Frame: From first dose to the date of the first documented response (up to approximately 34 months)
Population: Pre-specified for all treated participants in group A, B, and C only
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID)
Number analyzed (Participants) | 55 | 46 | 22
Percent of participants | 50.9 [37.1 to 64.6] | 45.7 [30.9 to 61.0] | 54.5 [32.2 to 75.6]

5. Secondary Outcome: Overall Survival for Participants With No Prior Systemic Therapy
Description: The time (in months) from first dosing until the date of death. For those participants who have not died, survival duration will be censored at the last date the participant was known to be alive.
Time Frame: From first dose to the date of death (up to approximately 34 months)
Population: Pre-specified for all treated participants in group A only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A (Brivanib 800 mg QD)
Number analyzed (Participants) | 55
Months | 9.95 [6.77 to 15.21]

6. Secondary Outcome: Overall Survival for Participants With One Prior Angiogenesis Inhibitor Therapy
Description: as for outcome 5
Time Frame: From first dose to the date of death (up to approximately 34 months)
Population: Pre-specified for all treated participants in group B and C only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group B (Brivanib 800 mg QD) | Group C (400 mg BID)
Number analyzed (Participants) | 46 | 22
Months | 9.79 [5.52 to 13.17] | 8.25 [6.83 to NA] — Insufficient number of events

7. Secondary Outcome: Progression Free Survival (PFS) Per Independent Response Review Committee (IRRC)
Description: The time (in months) from first dosing date to the date of progression per IRRC. Participants who die without a reported prior progression will be considered to have progressed on their date of death (as found in the BMS clinical database). Participants who did not progress or die will be censored on the date of their last tumor assessment. Participants who have only baseline tumor assessment will be censored on the first dosing date.
  Progression is defined as a 25% or more increase in the sum of all index lesion areas taking as reference the smallest sum recorded at or following baseline.
Time Frame: From first dose to the date of the first documented progression (up to approximately 34 months)
Population: Pre-specified for all treated participants in group A, B, and C only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID)
Number analyzed (Participants) | 55 | 46 | 22
Months | 2.69 [1.45 to 2.96] | 2.0 [1.41 to 3.91] | 2.96 [1.38 to 5.55]

8. Secondary Outcome: Time to Response Per Independent Response Review Committee (IRRC)
Description: The time from the first dose of study therapy until measurement criteria are first met for Partial response (PR) or complete response (CR), whichever is recorded first.
  Complete Response (CR): Disappearance of all known disease. Must be confirmed 4 or more weeks later.
  Partial Response (PR): A 50% or more decrease in the sum of all index lesion areas compared to the baseline sum and no unequivocal progression of existing non-index lesions. In addition, there can be no appearance of new lesions. Must be confirmed 4 or more weeks later.
Time Frame: From first dose to the date of the first documented response (up to approximately 34 months)
Population: Pre-specified for all treated participants in group A, B, and C only whose best response is either PR or CR
Measure: Median (Full Range); unit: Months
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD)
Number analyzed (Participants) | 4 | 2
Months | 10.4 [1.4 to 20.7] | 1.4 [1.4 to 1.4]

9. Secondary Outcome: Duration of Response Per Independent Response Review Committee (IRRC)
Description: Duration of response will be computed as from time measurement criteria are met for PR or CR until the date of documented progressive disease or death. Participants who neither relapse nor die will be censored on the date of their last tumor assessment. Progression is defined as a 25% or more increase in the sum of all index lesion areas taking as reference the smallest sum recorded at or following baseline.
  Complete Response (CR): Disappearance of all known disease. Must be confirmed 4 or more weeks later.
  Partial Response (PR): A 50% or more decrease in the sum of all index lesion areas compared to the baseline sum and no unequivocal progression of existing non-index lesions. In addition, there can be no appearance of new lesions. Must be confirmed 4 or more weeks later.
Time Frame: From first dose to the date of documented progressive disease or death (up to approximately 34 months)
Population: Pre-specified for all treated participants in group A, B, and C only whose best response is either PR or CR
Measure: Median (Full Range); unit: Months
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD)
Number analyzed (Participants) | 4 | 2
Months | 2.9 [1.4 to 20.7] | 4.2 [2.8 to 5.5]

10. Secondary Outcome: Change From Baseline to End of Treatment in FHSI-8 Total Score
Description: FHSI-8 (Functional Assessment of Cancer Therapy, Hepatobiliary, Symptom Index) was used to assess HCC-related symptoms. The FHSI-8 includes eight items representing HCC-related symptoms; each symptom is rated by participants on a scale of from 0 to 4. The FHSI-8 total score ranges in value from 0 to 32, with higher scores representing fewer symptoms and lower scores representing more symptoms.
Time Frame: Baseline and end of treatment (up to approximately 33 months)
Population: Pre-specified for all treated participants in group A, B, and C only with baseline and end of treatment measurements
Measure: Mean (Standard Deviation); unit: Change from baseline in FSHI-8 score
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID)
Number analyzed (Participants) | 38 | 35 | 18
Change from baseline in FSHI-8 score | -4.01 (8.37) | -2.40 (4.72) | -1.06 (6.98)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from participants first dose to their study completion (up to approximately 34 months). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 34 months)
Groups:
- Doxorubicin Cross-Over Participants: Participants who were randomized into the doxorubicin arm, prior to Amendment 7, and crossed-over to brivanib alaninate after disease progression (not failure of doxorubicin therapy due to toxicity alone), provided that they progressed either during doxorubicin therapy or after doxorubicin and no other therapy for HCC had been subsequently administered.
Arm/Group | Group A (Brivanib 800 mg QD) | Group B (Brivanib 800 mg QD) | Group C (400 mg BID) | Cohort D: Doxorubicin | Doxorubicin Cross-Over Participants
All-Cause Mortality (participants affected / at risk) | 39/55 | 37/46 | 13/22 | 4/14 | 3/6
Serious Adverse Events (participants affected / at risk) | 24/55 | 17/46 | 5/22 | 5/14 | 5/6
Other Adverse Events (participants affected / at risk) | 54/55 | 45/46 | 22/22 | 14/14 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Brivanib 800 mg QD) (N=55) | Group B (Brivanib 800 mg QD) (N=46) | Group C (400 mg BID) (N=22) | Cohort D: Doxorubicin (N=14) | Doxorubicin Cross-Over Participants (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0
Gait Disturbance (General disorders) | 2 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 2 | 0 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Gallbladder Disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 3 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Jaundice Hepatocellular (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Biliary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritoneal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Salmonella Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ammonia Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
International Normalised Ratio Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Platelet Count Decreased (Investigations) | 1 | 1 | 0 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 3 | 0 | 0 | 0
Hepatic Encephalopathy (Nervous system disorders) | 3 | 0 | 0 | 0 | 2
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Nephropathy Toxic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Renal Infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Venous Occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Brivanib 800 mg QD) (N=55) | Group B (Brivanib 800 mg QD) (N=46) | Group C (400 mg BID) (N=22) | Cohort D: Doxorubicin (N=14) | Doxorubicin Cross-Over Participants (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1 | 3 | 0 | 0
Left Ventricular Hypertrophy (Cardiac disorders) | 1 | 1 | 0 | 2 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 4 | 2 | 0 | 0 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Ventricular Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 5 | 7 | 4 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 4 | 2 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 7 | 5 | 3 | 3 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 9 | 6 | 3 | 0 | 1
Ascites (Gastrointestinal disorders) | 6 | 1 | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 9 | 10 | 5 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 23 | 19 | 8 | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 7 | 2 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 6 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 3 | 1 | 1 | 1
Faeces Discoloured (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 21 | 19 | 7 | 4 | 2
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 6 | 11 | 2 | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 16 | 14 | 7 | 0 | 0
Asthenia (General disorders) | 6 | 3 | 0 | 2 | 0
Chest Pain (General disorders) | 1 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 25 | 27 | 14 | 3 | 3
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 3 | 1 | 1 | 3 | 0
Oedema (General disorders) | 0 | 2 | 2 | 0 | 1
Oedema Peripheral (General disorders) | 11 | 2 | 5 | 3 | 1
Pain (General disorders) | 2 | 2 | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 4 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 7 | 3 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 7 | 4 | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 2 | 1 | 0 | 1 | 0
Ejection Fraction Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram St-T Change (Investigations) | 0 | 0 | 0 | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 2 | 3 | 0
Platelet Count Decreased (Investigations) | 1 | 4 | 3 | 3 | 0
Qrs Axis Abnormal (Investigations) | 2 | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 16 | 5 | 3 | 1 | 0
Weight Increased (Investigations) | 1 | 0 | 1 | 2 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 1 | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 22 | 25 | 8 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 5 | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 4 | 2 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 11 | 6 | 4 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 3 | 2 | 0 | 0
Headache (Nervous system disorders) | 10 | 11 | 1 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 2 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 1 | 0
Confusional State (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 4 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2 | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 4 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 8 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 1 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 6 | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 2 | 0 | 0
Hypertension (Vascular disorders) | 26 | 19 | 11 | 0 | 1
Venous Occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study protocol was amended to discontinue the doxorubicin arm, since doxorubicin was now considered an obsolete standard of care. The protocol was amended to add a third cohort of second-line participants receiving 400-mg brivanib alaninate BID for a total daily dose of 800 mg. The analyses for both cohorts are considered exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.